CLINICAL TRIAL: NCT05771168
Title: Observational Study for Patients Undergoing Surgery for Male Stress Urinary Incontinence
Brief Title: Surgery for Male Stress Urinary Incontinence
Acronym: SMUI
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Sacco Emilio, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 5094
Record Dates: First submitted 2023-02-03; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Male Stress Urinary Incontinence
Keywords: Urinary incontinence; Male incontinence; Post-prostatectomy incontinence; Radical prostatectomy; Male sling; Artificial urinary sphincter
MeSH Terms: conditions — Urinary Incontinence | interventions — Urinary Sphincter, Artificial; Suburethral Slings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AUS: Male patients undergoing surgery for stress urinary incontinence using artificial urinary sphincter (AUS)
  Interventions: Device: Artificial urinary sphincter
- Sling: Male patients undergoing surgery for stress urinary incontinence using slings
  Interventions: Device: Male sling

INTERVENTIONS:
Device: Artificial urinary sphincter — Implantation of peri-urethral artificial urinary sphincter
  Groups: AUS
Device: Male sling — Retrourethral implantation of male sling
  Groups: Sling

SUMMARY:
The purpose of this observational prospective study is to evaluate the success rate (cure plus improvement) of procedures for treatment of male stress urinary incontinence (artificial urinary sphincter or male slings) at 5 years of study follow-up and to determine other outcomes of surgical treatment for each of the devices and, to perform a prognostic factor analysis to identify clinical and surgical variables that correlate with (in)continence or revisions for each of the device subtypes. Cure is defined as urinary continence with no need for use of pads or the use of 1 light security pad; the improvement is defined as the reduction of≥ 50% of the number of pads with use of no more than two pads.

DETAILED DESCRIPTION:
Through the use of a prospective registry, the investigators will collect information on patient characteristics, including age (years), weight (kg), length (cm), previous urological surgeries and other surgeries in the pelvic area, radiotherapeutic treatment of the prostate, and other co-morbidities. Also, if applicable, 24h pad test and preoperative urodynamic results, presence of pre-operative urinary tract infections, and results of preoperative cystoscopy will be reported.

The surgical procedure for treatment of male stress urinary incontinence is according to standard practice. For artificial urinary sphincters, the date and time of surgery, surgeon name, time of shaving, presence of skin wounds, type of prosthesis, cuff location, cuff size, pressure regulating balloon, type of preoperative antibiotics, type of associated procedures will be reported. For slings, similar data will be reported, including type of sling and if there was a release of central tendon.

The patients will fill in the International Consultation on Incontinence Questionnaire (ICIQ) Urinary Incontinence (UI) Short Form (ICIQ-UI Questionnaire SF), the EuroQol Group Questionnaire (EQ-5D-5L) for the evaluation of the impact of incontinence on Quality of Life, and the Sexual Complaints Screener for Men (SCS-M), the Dyadic Adjustment Scale Italian version (DAS), the International Index of Erectile Function Questionnaire (IIEF-15) and the Hospital Anxiety and Depression Scale (HADS) questionnaire before the operation, at 12 weeks after surgery and at yearly intervals up to and including year 5. The results of questionnaires will be entered into the database.

ELIGIBILITY:
Inclusion Criteria:

* Male patients undergoing surgery for stress incontinence using medical devices such as AUS or sling
* Participant is willing and able to complete the questionnaires and give informed consent for participation in the study

Exclusion Criteria:

- Participant unable to complete the questionnaires and declining informed consent for participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patients undergoing surgery for treatment of stress urinary incontinence (AUS or male sling)
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Success rate (cure plus improvement) | 5-years after surgery
  Will be obtained through patient 24-hour pad use. Cure rate is defined as urinary continence with no need for use of pads or the use of 1 light security pad.

SECONDARY OUTCOMES:
Time being continent | 12-weeks, 12-months, 2-years, 3-years, 4-years, 5-years
  Interval being continent after surgery to the date of incontinence recurrence. Patients who die will be censored at time of death. Overall time of being continent will be presented using the Kaplan-Meier curve.
Time being revision-free | 12-weeks, 12-months, 2-years, 3-years, 4-years, 5-years
  Interval from the date of surgery to the date of revision.Patients who die will be censored at time of death. Overall time of being revision-free will be presented using the Kaplan-Meier curve.
Revision-free rate | 5-years after surgery
  Evaluation of revision-free rate at 5 years of study follow-up
Patient-reported quality of life | 12-weeks, 12-months, 2-years, 3-years, 4-years, 5-years
  The change in the results of quality of life questionnaires (EuroQol Group EQ-5D-5L) compared with baseline over time and correlations with the primary outcome. EuroQol Group EQ-5D-5L describe health state with 5 levels (level 1 indicating no problem, level 2 indicating slight problems, level 3 indicating moderate problems, level 4 indicating severe problems, level 5 indicating unable to/extreme problems) and with a scale numbered from 0 to 100 (100 means the best health you can imagine and 0 means the worst health you can imagine)
Post-operative general adverse events | 12-weeks, 12-months, 2-years, 3-years, 4-years, 5-years
  Post-operative general adverse events related to the surgical procedure or the sling/sphincter (e.g. urinary retention, scrotal hematoma, perineal pain, hematuria, or other general problems)
Post-operative specific adverse events | 12-weeks, 12-months, 2-years, 3-years, 4-years, 5-years
  Post-operative specific adverse events related to the surgical procedure or the sling/sphincter (e.g. pump/reservoir/cuff failure, erosion of the device through the skin or urethra)

CONTACTS AND LOCATIONS:
Locations (1):
- Università Cattolica del Sacro Cuore, Fondazione Policlinico Agostino Gemelli, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No